CLINICAL TRIAL: NCT03505632
Title: Low Positive End Expiratory Pressure With Alveolar Recruitment Maneveurs Versus High Positive End Expiratory Pressure as Lung Protective Strategy in Laparoscopic Bariatric Surgeries
Brief Title: High Versus Low Positive End Expiratory Pressure With Alveolar Recruitment Maneuver in Laparoscopic Bariatric Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mahmoud Othman, professor of Anesthesia and surgical ICU, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MD/16.3.24
Record Dates: First submitted 2018-04-05; First posted 2018-04-23 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Anesthesia

STUDY DESIGN:
Intervention Model Description: Mechanical ventilation with either recruitment maneuver and low PEEP versus conventional mechanical ventilation and high PEEP
Who Masked: Participant, Outcomes Assessor
Masking Description: This study is double blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Recruitment with low PEEP (Experimental): Recruitment maneuver ( RM) will carried out during 2 minutes with increasing PEEP in stepwise manner.PEEP increase from 5 to 10 cmH2O (3 breaths),then to 15 cm H2O (3 breaths), PEEP to 20 cmH2O (10 breaths).Then decrease by 5 cmH2O every 3 breaths till back to preset PEEP 5 cmH2O .Recruitment carried out at the following times: post intubation(T1) , after insuflation(T2) ,after desuflation (T3) and before extubation(T4) . The peak airway pressure should not exceed 40cmH2O .
  Interventions: Device: Recruitment with low PEEP
- High PEEP without RM (Active Comparator): Patients will receive from the start during anesthesia high PEEP (15 cmH2O) with maintaining the peak airway pressure below 40 cm H2O.
  Monitoring times: after intubation(T1), post-insufflation(T2), after desuflation (T3) and before extubation(T4).
  Interventions: Device: High PEEP without RM

INTERVENTIONS:
Device: Recruitment with low PEEP — Volume controlled ventilation with TV 6-8 ml/PBW . RR adjusted to keep the EtCO2 35-40 mmHg. I/E ratio1:2 and FiO2 0.40.Patients will receive PEEP of 5cmH2O. RM will be done by increasing the PEEP in stepwise manner. First PEEP increase to 10 cmH2O (3 breaths),then to 15 cm H2O (3 breaths) and finally PEEP raise to 20 cmH2O (10 breaths).Then PEEP decrease by 5 cmH2O increments every (3 breaths) until back to PEEP 5 cmH2O. RM will take 2 minutes. RM will be carried out at the following times: post intubation(T1) , after peritoneal insuflation(T2) ,after desuflation (T3) and before extubation(T4) . The peak airway pressure should not exceed 40 cmH2O. Monitoring of the following parameters :Dynamic lung compliance ,Horowitz index ,dead space and driving pressure .
  Other Names: Low PEEP + RM
  Arms: Recruitment with low PEEP
Device: High PEEP without RM — Volume controlled ventilation will carried out with tidal volume 6-8 ml/kg for predicted body weight. The PBW calculated according to the formula : 50 + 0.91 × {height (cm)-152.4} for men and 45.5 + 0.91 × {height (cm) - 152.4} for women. The respiratory rate adjusted to keep the EtCO2= 35-40 mmHg. The inspiratory to expiratory ratio (I:E ratio) 1:2 and FiO2 0.40.Patients will receive high PEEP of 15cmH2O from the start and continue all through the procedure . Monitoring of dynamic lung compliance,Horowitz index,dead space and driving pressure will be carried out at the following times: post intubation(T1) , after peritoneal insuflation(T2) ,after desuflation (T3) and before extubation(T4) . The peak airway pressure should not exceed 40cmH2O.
  Other Names: High PEEP
  Arms: High PEEP without RM

SUMMARY:
For the patients undergoing laparoscopic bariatric surgery, application of low (PEEP) with frequent alveolar recruitment maneuver could be beneficial and superior to conventional ventilation with a high (PEEP) in improving lung compliance, better oxygenation and less dead space .This hypothesis could be achieved by minimizing the expected lung atelectasis during anesthesia for this particular kind of laparoscopic surgery without any haemodynamics alterations.This trial was designed to study the effects of alveolar recruitment strategy with low PEEP versus conventional mechanical ventilation with higher PEEP on the patients undergoing laparoscopic bariatric surgeries. The primary end point of the study will be the achievement of the highest dynamic lung compliance (Cdyn). Improvement of intraoperative oxygenation (Pao2/Fio2) and achievement of a lower dead space ratio (vd/vt), with stable intraoperative haemodynamics will be considered as secondary outcome

DETAILED DESCRIPTION:
The use of a alveolar recruitment maneuver(RM) effectively increases end expiratory lung volume and reopens lung atelectasis during anesthesia and reproduces better oxygenation for surgical obese patients .Alveolar recruitment maneuver with PEEP could decreases atelectasis and improved oxygenation in obese surgical patients .This concept indicate that the maintenance of low PEEP after multiple alveolar recruitment maneuver during anesthesia may improve its benefits without complications. Patients will randomly divided by computerized randomization sequence method into two groups (30 patients in each study group):

Both groups receive volume controlled ventilation, tidal volume was 6-8 ml/kg for predicted body weight. The PBW calculated according to a formula: 50 + 0.91 × {height (cm)-152.4} for men and 45.5 + 0.91 × {height (cm) - 152.4} for women. The respiratory rate was adjusted to keep the EtCO2= 35-40 mmHg. The inspiratory to expiratory ratio (I:E ratio) was 1:2 and the FiO2 was 0.40.

Low PEEP+RM group: Patients receive PEEP of 5cmH2O. Recruitment maneuver ( RM) will be done by increasing the PEEP in stepwise manner. First PEEP was increased to 10 cmH2O (3 breaths),then to 15 cm H2O (3 breaths).Finally, PEEP was raised to 20 cmH2O (10 breaths).Then decreased for 15cmH2O for (3 breaths),10cmH2O for(3 breaths), and finally returned back to original PEEP 5 cmH2O.The total procedure took 2 min. Recruitment will be carried out at the following times: post intubation(T1) , after peritoneal insuflation(T2) ,after desuflation (T3) and before extubation(T4) . The peak airway pressure should not exceed 40cmH2O.

High PEEP group: Patients receive throughout ventilation 15 cm H2O PEEP with maintaining the peak airway pressure below 40 cm H2O.

Monitoring :after intubation(T1), post-insufflation(T2), after disinflation (T3) and before extubation(T4) for the fillowoing.1--Minute volume ,respiratory rate and tidal volume 2-Arterial blood gas( PaO2, PaCO2,pH).3-Hemodynamics : heart rate and invasive arterial blood pressure.4-Calculated dynamic Lung compliance by equation: T V/peak airway pressure- PEEP .5-calculated driving pressure by equation: Pplat-PEEP.6-Calculated dead space ratio (VD/VT) by equation :PaCO2-ETCO2)/ PaCO2.

Rescue strategies:

A) Intraoperative hypoxemia (SpO2≤92%): In both groups ,rescue primarily will be performed by an increase in FiO2 by 0.1 till reaching oxygen (100% ) .If failed and hypoxia persist a recruitment maneuver will be carried out with stepwise incremental PEEP irrespective of the group allocation.

The time of the event of hypoxia and its management will be recorded.

B) Intraoperative hypotension (systolic blood pressure <90 mmHg):

1. Abort any recruitment maneuver in low PEEP+ RM group.
2. Gradual decrease PEEP by 5 cmH2O in stepwise manner in higher PEEP group.
3. Give 500 ml bolus colloid and correct fluid status with blood transfusion if indicated.
4. Noradrenalin infusion as last resort

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) physical status II and III.
2. Patients included in the study having body mass index ≥35kg/m2.
3. Both genders.
4. Age ≥ 20 years old.

Exclusion Criteria:

1. Major cardiovascular diseases (heart failure and ejection fraction below 40%).
2. Sever obstructive pulmonary diseases (FEV1 < 50 and FVC < 50)
3. Hepatic and renal impairment.
4. Younger than 20 years old.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Dynamic lung compliance | During intra-operative mechanical ventilation
  To achieve nearly 20% increase in dynamic lung compliance (Cdyn) during anesthesia for obese patients undergoing bariatric surgery.

SECONDARY OUTCOMES:
Horowitz ratio | During mechanical ventilation
  Improvement of intraoperative oxygenation with Horowitz ratio (Pao2/Fio2) more than 350.
Alveolar dead space ratio | During mechanical ventilation
  Achievement of the least alveolar dead space ratio (vd/vt).
Systolic blood pressure | During mechanical ventilation
  Maintain systolic blood pressure above 100 mmHg.
Diastolic blood pressure | During mechanical ventilation
  Maintain diastolic blood pressure above 50 mmHg.
Mean blood pressure | During mechanical ventilation
  Maintain mean blood pressure above 65 mmHg.
Heart rate | During mechanical ventilation
  Maintain heart rate within the range of 60-90 (bpm ).
Analgesia | postoperative time for 24 hours
  postoperative visual analogue score less than 4.
Atelectasis | postoperative time for 24 hours
  Chest X-ray for evidences of atelectasis

CONTACTS AND LOCATIONS:
Overall Officials: Amgad A Zaghloul, MD, Study Chair — Mansoura University; Ahmed M Farid, MD, Study Chair — Mansoura University
Locations (1):
- Mansoura faculty of medicine, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
No available other researchers